CLINICAL TRIAL: NCT07346053
Title: CHRONO-EVP: Time-of-day Dependent Administration of Enfortumab Vedotin and Pembrolizumab (EV/P) in Advanced Bladder Cancer
Brief Title: The Impact of Time-of-day Administration of EV/P on Objective Response Rate in Adults With Advanced Bladder Cancer
Acronym: Chrono-EVP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guliz Ozgun (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor-Investigator, Guliz Ozgun, Medical Oncologist, Principal Investigator, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chrono-EVP
Record Dates: First submitted 2025-12-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Bladder Cancer
Keywords: time-of-day administration; chronotherapy; advanced bladder cancer; circadian rhythm; enfortumab vedotin and pembrolizumab (EV/P); urothelial cancer; chronoimmunotherapy
MeSH Terms: interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled trial designed to evaluate the effects of timing of standard-of-care (SOC) treatment administration on patient outcomes. Participants will be randomly assigned to receive SOC enfortumab vedotin and pembrolizumab (EV/P) either in the morning or in the afternoon, with no additional interventions planned. Patients will be scheduled for treatments at the same time for the first four cycles, with a ±1 hour flexibility, to minimize the impact of timing as a confounding factor in the analyses. To preserve the immune priming effect, which is most pronounced during the initial treatment period, infusion timing will be strictly enforced during the first four cycles. After this period, patients will be allowed to have a flexible schedule. Treatment will be initiated in accordance with the standard of care, with no additional interventions planned. The trial is open-label and not blinded due to the nature of the intervention (timing of treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Morning EV/P Treatment (Active Comparator): Participants will receive standard-of-care therapy (Ev/P) administered in the morning (before 11:30am).
  Interventions: Drug: enfortumab vedotin and pembrolizumab (EV/P)
- Arm B: Afternoon EV/P Treatment (Active Comparator): Participants will receive standard-of-care therapy (EV/P) administered in the afternoon (after 1:30pm).
  Interventions: Drug: enfortumab vedotin and pembrolizumab (EV/P)

INTERVENTIONS:
Drug: enfortumab vedotin and pembrolizumab (EV/P) — Participants will receive EV/P as part of their standard-of-care therapy administered either in the morning (Arm A) or afternoon (Arm B), as determined by randomization.

SUMMARY:
The goal of this clinical trial is to learn if the timing of treatments plays a role in how effective the standard-of-care drugs enfortumab vedotin and pembrolizumab (EV/P) works to treat adults with advanced bladder cancer. The trial will also learn if time-of-day reduces EV/P side-effects.

Researchers will compare EV/P given in the morning (before 11:30am) vs in the afternoon (after 1:30pm), to see if circadian rhythm effects how EV/P works to treat advanced bladder cancer.

Participants will be randomized in Arm A or Arm B to receive drugs EV/P either in the morning (Arm A) or afternoon (Arm B) as part of their standard-of-care treatment for advanced bladder cancer. Participants will:

* Visit the clinic either in the morning (Arm A) or afternoon (Arm B) to receive EV/P treatment as part of their regular medical care for advanced bladder cancer
* Frequency of visits will follow standard-of-care guidelines
* Participants will be followed-up by the study team for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following inclusion criteria to be eligible for participation in this trial:

  1. Age 18 or older
  2. Able to provide informed consent
  3. Histologically confirmed advanced urothelial cancer
  4. Eligible for standard-of-care EV/P regimen
  5. Measurable disease per RECIST 1.1
  6. ECOG performance status 0-2
  7. Ability to adhere to scheduled infusion times (Before 11:30 a.m. or after 1:30 pm) Waivers to the inclusion criteria will NOT be allowed.

Exclusion Criteria:

* Participants who meet any of following exclusion criteria will not be eligible for participation in this trial:

  1. Non-urothelial histology or mixed histology with predominant non-urothelial components
  2. Concurrent malignancy requiring active systemic therapy, unless disease-free for at least 2 years
  3. Inability to comply with protocol-specified infusion timing for at least the first 3 months
  4. Night shift workers
  5. Clinical evidence of new or enlarging brain metastasis or carcinomatous meningitis
  6. Known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial
  7. Patients who have traveled across ≥2 time zones within the past 14 days prior to randomization will be excluded, due to potential disruption of circadian rhythms (jet lag), which may affect chronotherapy-related endpoints.
  8. Patients with a clinically diagnosed sleep disorder, including but not limited to insomnia, obstructive sleep apnea, restless leg syndrome, or circadian rhythm sleep-wake disorders, that is moderate to severe, untreated, or poorly controlled, will be excluded.

Waivers to the exclusion criteria will NOT be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate in in time-of-day administration of EV/P treatment | From enrollment to end of follow-up at 24-months.
  Objective response rate (ORR) will be determined by proportion of patients achieving a complete or partial response as assessed by RECIST v1.1 criteria, confirmed by central review or investigator assessment. Tumor assessments will be performed as standard of care (typically every 12 weeks), and best overall response prior to disease progression will be used for ORR determination.

SECONDARY OUTCOMES:
Evaluate Progression-Free Survival in time-of-day administration of EV/P | From enrollment to end of follow-up at 24-months.
  Progression-free Survival (PFS) will be determined by time of randomization to radiographic progression or death from any cause, whichever occurs first.
Assess Overall-Survival in time-of-day administration of EV/P | From enrollment to the end of follow-up at 24-months.
  Overall-survival (OS) is defined as the time from randomization to death from any cause. The analysis will compare OS curves between study arms and estimate 2-year OS rates for each group.
Evaluate the Time-to-Treatment Failure in time-of-day administration of EV/P | From enrollment to the end of follow-up at 24-months.
  Time to treatment failure (TTF) is determined by assessing time from treatment initiation to treatment discontinuation for any reason, including disease progression, unacceptable toxicity, patient withdrawal, or death, capturing both treatment efficacy and tolerability.
Assess quantitative changes in ctDNA Kinetics of time-of-day administration of EV/P | Baseline, 3 weeks, and 12-weeks.
  Quantitative changes in circulating tumour DNA (ctDNA) levels will be collected and measured at baseline, post-cycle 1 (~3 weeks), and at post-cycle 4 (~12 weeks) at first radiographic assessment, with correlation to response and survival outcomes.
Assess treatment-related tolerability and toxicity differences | From enrollment to the end of follow-up at 24-months.
  Differences in steroid use (yes/no) for the management of treatment-related toxicity, treatment interruptions (yes/no) due to treatment-related toxicity, and treatment discontinuations (yes/no) due to treatment-related toxicity will be used as surrogate safety outcomes, as comprehensive adverse event documentation is beyond the scope of this pragmatic clinical trial. The study seeks to determine whether treatment administration at a predefined time of day is associated with differences in the need for toxicity-related clinical interventions. Given that the relevant adverse events are well characterized in the existing literature, the focus of this study is on comparative safety between groups using these surrogate measures rather than on detailed characterization of individual adverse events.
Immune Profiling | At 4 time points: Baseline, 1-day post first cycle of treatment, 3 weeks into treatment and 12 weeks into treatment
  Immune cell populations will be characterized from the blood samples at baseline (prior to treatment initiation) and at three predefined time points during therapy: 1 day after treatment initiation, 3 weeks into treatment, and 12 weeks into treatment. Cytometry by time-of-flight (CyTOF) will be used to comprehensively profile immune cell populations allowing for high-dimensional assessment of immune cell composition and activation states across treatment timing groups.
Bulk RNA sequencing (RNA-seq) | At 4 time points: Baseline, 1-day post first cycle of treatment, 3 weeks into treatment and 12 weeks into treatment
  Bulk RNA sequencing (RNA-seq) will be performed to comprehensively characterize global gene expression profiles and to evaluate time-of-day-associated differences in immune-related transcriptional signatures. This approach will enable the identification of circadian variation in gene expression and provide insight into temporal regulation of immune pathways in response to treatment.
Cytokine and chemokine analyses | At 4 time points: Baseline, 1-day post first cycle of treatment, 3 weeks into treatment and 12 weeks into treatment
  Plasma will be isolated for cytokine and chemokine analyses to assess systemic immune signaling and inflammatory profiles. Quantitative evaluation of circulating cytokines and chemokines will provide insight into treatment- and time-dependent changes in immune activation, inflammation, and immune regulation, complementing cellular and transcriptional immune profiling.
Circulating Tumor DNA (ctDNA) Analyses | At 3 time points: Baseline, 3 weeks into treatment and 12 weeks into treatment
  Circulating tumor DNA (ctDNA) analyses will be performed on plasma samples collected at baseline (prior to treatment initiation), 3 weeks into treatment, and 12 weeks into treatment. ctDNA dynamics will be evaluated to assess molecular response to therapy, including changes in ctDNA levels and ctDNA clearance rates over time. Comparisons will be made between treatment administration at different times of day to determine whether timing of therapy is associated with differences in ctDNA kinetics, clearance rates, and early molecular response.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - BC Cancer - Abbotsford, Abbotsford, British Columbia
  - BC Cancer - Kelowna (Sindi Ahluwalia Hawkins Centre), Kelowna, British Columbia
  - BC Cancer - Surrey, Surrey, British Columbia
  - BC Cancer - Vancouver Cancer Centre, Vancouver, British Columbia
  - BC Cancer - Victoria, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang C, Zeng Q, Gul ZM, Wang S, Pick R, Cheng P, Bill R, Wu Y, Naulaerts S, Barnoud C, Hsueh PC, Moller SH, Cenerenti M, Sun M, Su Z, Jemelin S, Petrenko V, Dibner C, Hugues S, Jandus C, Li Z, Michielin O, Ho PC, Garg AD, Simonetta F, Pittet MJ, Scheiermann C. Circadian tumor infiltration and function of CD8+ T cells dictate immunotherapy efficacy. Cell. 2024 May 23;187(11):2690-2702.e17. doi: 10.1016/j.cell.2024.04.015. Epub 2024 May 8. PMID 38723627
- [Background] Fortin BM, Pfeiffer SM, Insua-Rodriguez J, Alshetaiwi H, Moshensky A, Song WA, Mahieu AL, Chun SK, Lewis AN, Hsu A, Adam I, Eng OS, Pannunzio NR, Seldin MM, Marazzi I, Marangoni F, Lawson DA, Kessenbrock K, Masri S. Circadian control of tumor immunosuppression affects efficacy of immune checkpoint blockade. Nat Immunol. 2024 Jul;25(7):1257-1269. doi: 10.1038/s41590-024-01859-0. Epub 2024 May 28. PMID 38806707
- [Background] Lee Y. Roles of circadian clocks in cancer pathogenesis and treatment. Exp Mol Med. 2021 Oct;53(10):1529-1538. doi: 10.1038/s12276-021-00681-0. Epub 2021 Oct 7. PMID 34615982
- [Background] Goncalves L, Guedes H, Fortuna AR, Lemos T, Gramaca J, Mourao N, Cunha G, Pichel R, Simoes P, Luis JA, Freitas R, Dunoes I, Spencer AS, Marinho J, Costa L. Avelumab Maintenance Therapy in Advanced Urothelial Carcinoma: Implications of Timing and Treatment Sequencing. Cancers (Basel). 2025 Mar 6;17(5):898. doi: 10.3390/cancers17050898. PMID 40075745
- [Background] Giacchetti S, Bjarnason G, Garufi C, Genet D, Iacobelli S, Tampellini M, Smaaland R, Focan C, Coudert B, Humblet Y, Canon JL, Adenis A, Lo Re G, Carvalho C, Schueller J, Anciaux N, Lentz MA, Baron B, Gorlia T, Levi F; European Organisation for Research and Treatment of Cancer Chronotherapy Group. Phase III trial comparing 4-day chronomodulated therapy versus 2-day conventional delivery of fluorouracil, leucovorin, and oxaliplatin as first-line chemotherapy of metastatic colorectal cancer: the European Organisation for Research and Treatment of Cancer Chronotherapy Group. J Clin Oncol. 2006 Aug 1;24(22):3562-9. doi: 10.1200/JCO.2006.06.1440. PMID 16877722
- [Background] Levi F, Okyar A, Dulong S, Innominato PF, Clairambault J. Circadian timing in cancer treatments. Annu Rev Pharmacol Toxicol. 2010;50:377-421. doi: 10.1146/annurev.pharmtox.48.113006.094626. PMID 20055686
- [Background] Powles T, Valderrama BP, Gupta S, Bedke J, Kikuchi E, Hoffman-Censits J, Iyer G, Vulsteke C, Park SH, Shin SJ, Castellano D, Fornarini G, Li JR, Gumus M, Mar N, Loriot Y, Flechon A, Duran I, Drakaki A, Narayanan S, Yu X, Gorla S, Homet Moreno B, van der Heijden MS; EV-302 Trial Investigators. Enfortumab Vedotin and Pembrolizumab in Untreated Advanced Urothelial Cancer. N Engl J Med. 2024 Mar 7;390(10):875-888. doi: 10.1056/NEJMoa2312117. PMID 38446675